CLINICAL TRIAL: NCT00908648
Title: The Impact of Narrow Band Imaging in Screening Colonoscopy: a Randomized Controlled Trial.
Brief Title: The Use of Narrow Band Imaging in Screening Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Vittorio Terruzzi, MD, Valduce Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NBI-01
Record Dates: First submitted 2009-01-22; First posted 2009-05-27 (Estimated); Results first posted 2009-05-27 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-03

CONDITIONS: Colonoscopy
Keywords: screening colonoscopy; narrow band imaging
MeSH Terms: interventions — Narrow Band Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): standard white light
- 2 (Experimental): Narrow Band Imaging
  Interventions: Procedure: Narrow Band Imaging

INTERVENTIONS:
Procedure: Narrow Band Imaging — Narrow Band Imaging
  Arms: 2

SUMMARY:
Narrow band imaging (NBI) is an imaging technique that allows a better definition of capillary pattern and improves the contrast between adenomas and the surrounding mucosa. Conflicting data exist on the ability of NBI in to improve detection of colonic neoplasm; the impact of NBI is being tested in several screening scenarios. The investigators evaluated whether the routine use of NBI, compared to white light (WL), during the withdrawal phase of screening colonoscopy improved adenoma detection.

ELIGIBILITY:
Inclusion Criteria:

* 50-69 year-old asymptomatic subjects at average-risk of CRC
* positive FOBT participating in a national mass-screening program and referred for colonoscopy

Exclusion Criteria:

* ongoing anticoagulation therapy
* inadequate bowel cleansing
* incomplete colonoscopy
* refusing to participate

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2007-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

REFERENCES:
- [Background] Machida H, Sano Y, Hamamoto Y, Muto M, Kozu T, Tajiri H, Yoshida S. Narrow-band imaging in the diagnosis of colorectal mucosal lesions: a pilot study. Endoscopy. 2004 Dec;36(12):1094-8. doi: 10.1055/s-2004-826040. PMID 15578301
- [Background] Chiu HM, Chang CY, Chen CC, Lee YC, Wu MS, Lin JT, Shun CT, Wang HP. A prospective comparative study of narrow-band imaging, chromoendoscopy, and conventional colonoscopy in the diagnosis of colorectal neoplasia. Gut. 2007 Mar;56(3):373-9. doi: 10.1136/gut.2006.099614. Epub 2006 Sep 27. PMID 17005766

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Gastroenterology Unit November 2007 - April 2008
Pre-assignment Details: Patients undergoing incomplete procedure for inadequate bowel cleansing or failure to reach the cecum were excluded from randomization
Groups:
- Standard White Light: use of standard white light during the withdrawal phase of colonoscopy
- Narrow Band Imaging: use of narrow band imaging during the withdrawal phase of colonoscopy
Period: Overall Study
Arm/Group | Standard White Light | Narrow Band Imaging
Started | 108 | 103
Completed | 108 | 103
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard White Light | Narrow Band Imaging | Total
Number analyzed (Participants) | 108 | 103 | 211
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 90 | 88 | 178
  >=65 years | 18 | 15 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (5.8) | 59.6 (5.3) | 60.8 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 47 | 94
  Male | 61 | 56 | 117

OUTCOME MEASURES:

1. Primary Outcome: Adenoma Detection
Description: Detection of adenoma, defined as the number of patients with > 1 adenoma, under White Light or NBI visualization
Time Frame: duration of colonoscopy procedure
Measure: Number; unit: participants
Arm/Group | Standard White Light | Narrow Band Imaging
Number analyzed (Participants) | 108 | 103
participants | 63 | 59

2. Secondary Outcome: Detection of Flat and/or Depressed Adenomas
Description: number of patients with at least 1 flat and/or depressed adenoma
Time Frame: duration of colonoscopy procedure
Measure: Number; unit: participants
Arm/Group | Standard White Light | Narrow Band Imaging
Number analyzed (Participants) | 108 | 103
participants | 10 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No